CLINICAL TRIAL: NCT03029286
Title: ENGAGED 2 Study: Experiences With Mammography Screening and Breast Density 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: Kaiser Permanente (Other)
Responsible Party: Principal Investigator, Suzanne C. O'Neill, Associate Professor, Georgetown University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2015-0687
Record Dates: First submitted 2017-01-18; First posted 2017-01-24 (Estimated); Results first posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Breast Density; Breast Cancer Female
Keywords: Breast Cancer; Breast Density
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized Web Intervention Arm (Experimental): Women will be assigned to view a tailored website featuring their personalized risk information for breast cancer related to breast density and other factors.
  Interventions: Behavioral: Personalized Web Intervention Arm
- Usual Care Arm (Active Comparator): Women will be assigned to view a website that will take them to the American Cancer Society website to view general risk information for breast cancer related to breast density.
  Interventions: Behavioral: Usual Care Arm

INTERVENTIONS:
Behavioral: Usual Care Arm — Health information provided by the American Cancer Society Website
  Arms: Usual Care Arm
Behavioral: Personalized Web Intervention Arm — Women will be assigned to view a tailored website featuring their personalized risk information for breast cancer related to breast density and other factors.
  Arms: Personalized Web Intervention Arm

SUMMARY:
This trial will test a decision support web based intervention for women at increased risk for breast cancer due to breast density and other risk factors (age, race/ethnicity, family history of breast cancer, history of prior breast biopsies), and to consider MRI and/or chemoprevention to manage their breast cancer risk.

DETAILED DESCRIPTION:
Along with better-known risk factors such as family history having dense breasts is one of the strongest breast cancer risk factors. Extremely dense breast tissue affects about 10% of women, with an additional third having heterogeneously dense breasts. Women in these categories have 3-6 times the risk of breast cancer as compared to women with least density. Although breast density is measured on routine screening mammograms, it is not typically communicated to patients. This is changing as a result of legal mandates and approaches need to be tested to effectively integrate this clinical information in care. Therefore,we have developed an intervention to support decision making about cancer risk management (MRI and chemoprevention) for women at clinically elevated risk using a web-based intervention that will evaluate the efficacy of a web based intervention with personalized risk information communication versus usual care.

ELIGIBILITY:
Inclusion Criteria:

* Women, aged 40-69
* Enrolled at Group Health
* Have had a negative mammogram as part of their routine care
* Either (a) an intermediate 5-year risk (>1.67%-2.49%) and extremely dense breasts or (b) a high 5-year risk (≥2.50%) and either heterogeneously dense or extremely dense breasts utilizing the Breast Cancer Surveillance Consortium Risk Calculator (http://tools.bcsc-scc.org/BC5yearRisk/)
* Women must also have a valid email address.

Exclusion Criteria:

* Not able to speak and read English
* History of LCIS
* Prior cancer diagnosis (including DCIS)
* Known BRCA1/2 family mutation, or previous receipt of cancer genetic counseling
* Do not want to be contacted for research
* Have previously participated in intervention development activities
* Dis-enrolled from health plan between mammogram and start of recruitment.

Ages: 40 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 995 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne C O'Neill, PhD, Principal Investigator — Georgetown University/Lombardi Comprehensive Cancer Center; Karen Wernli, PhD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Washington Health Research Institute, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Knerr S, Wernli KJ, Leppig K, Ehrlich K, Graham AL, Farrell D, Evans C, Luta G, Schwartz MD, O'Neill SC. A web-based personalized risk communication and decision-making tool for women with dense breasts: Design and methods of a randomized controlled trial within an integrated health care system. Contemp Clin Trials. 2017 May;56:25-33. doi: 10.1016/j.cct.2017.02.009. Epub 2017 Feb 28. PMID 28257920
- [Result] Mahorter SS, Knerr S, Bowles EJA, Wernli KJ, Gao H, Schwartz MD, O'Neill SC. Prior breast density awareness, knowledge, and communication in a health system-embedded behavioral intervention trial. Cancer. 2020 Apr 15;126(8):1614-1621. doi: 10.1002/cncr.32711. Epub 2020 Jan 24. PMID 31977078
- [Result] Wernli KJ, Bowles EA, Knerr S, Leppig KA, Ehrlich K, Gao H, Schwartz MD, O'Neill SC. Characteristics Associated with Participation in ENGAGED 2 - A Web-based Breast Cancer Risk Communication and Decision Support Trial. Perm J. 2020 Dec;24:1-4. doi: 10.7812/TPP/19.205. PMID 33482952
- [Result] Wernli KJ, Knerr S, Li T, Leppig K, Ehrlich K, Farrell D, Gao H, Bowles EJA, Graham AL, Luta G, Jayasekera J, Mandelblatt JS, Schwartz MD, O'Neill SC. Effect of Personalized Breast Cancer Risk Tool on Chemoprevention and Breast Imaging: ENGAGED-2 Trial. JNCI Cancer Spectr. 2021 Jan 14;5(1):pkaa114. doi: 10.1093/jncics/pkaa114. eCollection 2021 Feb. PMID 33554037
- [Result] Bowles EJA, O'Neill SC, Li T, Knerr S, Mandelblatt JS, Schwartz MD, Jayasekera J, Leppig K, Ehrlich K, Farrell D, Gao H, Graham AL, Luta G, Wernli KJ. Effect of a Randomized Trial of a Web-Based Intervention on Patient-Provider Communication About Breast Density. J Womens Health (Larchmt). 2021 Nov;30(11):1529-1537. doi: 10.1089/jwh.2021.0053. Epub 2021 Sep 28. PMID 34582721
- [Result] Conley CC, Wernli KJ, Knerr S, Li T, Leppig K, Ehrlich K, Farrell D, Gao H, Bowles EJA, Graham AL, Luta G, Jayasekera J, Mandelblatt JS, Schwartz MD, O'Neill SC. Using Protection Motivation Theory to Predict Intentions for Breast Cancer Risk Management: Intervention Mechanisms from a Randomized Controlled Trial. J Cancer Educ. 2023 Feb;38(1):292-300. doi: 10.1007/s13187-021-02114-y. Epub 2021 Nov 23. PMID 34813048
- [Derived] Wernli KJ, Smith RE, Henderson LM, Zhao W, Durham DD, Schifferdecker K, Kaplan C, Buist DSM, Kerlikowske K, Miglioretti DL, Onega T, Alsheik NH, Sprague BL, Jackson-Nefertiti G, Budesky J, Johnson D, Tosteson ANA. Decision quality and regret with treatment decisions in women with breast cancer: Pre-operative breast MRI and breast density. Breast Cancer Res Treat. 2022 Aug;194(3):607-616. doi: 10.1007/s10549-022-06648-7. Epub 2022 Jun 20. PMID 35723793

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Personalized Web Intervention Arm | Usual Care Arm
Started | 492 | 503
Completed | 492 | 503
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Personalized Web Intervention Arm | Usual Care Arm | Total
Number analyzed (Participants) | 492 | 503 | 995
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.8 (5.02) | 61.9 (5.15) | 61.8 (5.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 492 | 503 | 995
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 9 | 5 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 10 | 19
  White | 465 | 478 | 943
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 8 | 8 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 8 | 16
  Not Hispanic or Latino | 484 | 495 | 979
  Unknown or Not Reported | 0 | 0 | 0
Distress related to cancer risk [Mean (Standard Deviation); unit: Distress thermometer (0-10)] — Distress was measured with the item, "Please choose the number (from 0-10) that best describes how much distress you have been experiencing related to your cancer risk in the past week including today, from 0 (no distress) to 10 (extreme distress).
  Distress thermometer (0-10) | 0.29 (1.08) | 0.21 (1.05) | 0.25 (1.06)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Taking Chemoprevention at 12 Months
Description: Number of Participants who initiated chemoprevention is measured as receipt of any prescription for tamoxifen or raloxifene, based on health plan pharmacy data at any time from consent through 12 months.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Personalized Web Intervention Arm | Usual Care Arm
Number analyzed (Participants) | 492 | 503
Participants | 1 | 1

2. Secondary Outcome: Distress Related to Cancer Risk
Description: Distress was measured with the item, "Please choose the number (from 0-10) that best describes how much distress you have been experiencing related to your cancer risk in the past week including today, from 0 (no distress) to 10 (extreme distress)."
Time Frame: 6 weeks and 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Personalized Web Intervention Arm | Usual Care Arm
Number analyzed (Participants) | 492 | 503
score on a scale
  Distress at 6 weeks | 0.72 (1.66) | 0.61 (1.51)
  Distress at 12 months | 0.36 (1.13) | 0.47 (1.34)

3. Secondary Outcome: Number of Participants Receiving Breast MRI
Description: Number of participants receiving breast MRI was assessed using EHR data on receipt of breast imaging within network or claims data from outside imaging facilities.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Personalized Web Intervention Arm | Usual Care Arm
Number analyzed (Participants) | 492 | 503
Participants | 16 | 3

ADVERSE EVENTS:
Time Frame: Participants could report any and all issues to the study team, from enrollment and consent through the 12 month survey.
Arm/Group | Personalized Web Intervention Arm | Usual Care Arm
All-Cause Mortality (participants affected / at risk) | 0/492 | 0/503
Serious Adverse Events (participants affected / at risk) | 0/492 | 0/503
Other Adverse Events (participants affected / at risk) | 0/492 | 0/503

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-08): https://cdn.clinicaltrials.gov/large-docs/86/NCT03029286/Prot_SAP_000.pdf